CLINICAL TRIAL: NCT04738851
Title: ARTHEMIRS: Assessment of Brain Activation During Different Mirror Therapy Tasks Using fNIRS Technology
Brief Title: Study of Cerebral Activation During Different Rehabilitation Tasks in Mirror Therapy in Healthy Subjects
Acronym: ARTHEMIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO 2020-14
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: mirror therapy; near infrared spectroscopy; cerebral activation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental): Virtual mirror therapy task : TMV Classic mirror therapy task : TMC Control task :TC
  Interventions: Other: Therapy Mirror task

INTERVENTIONS:
Other: Therapy Mirror task — The protocol has 3 conditions:
  * A virtual TM task (TMV
  * A classic TM task (TMC)
  * A control task (TC)
  The order of the 3 conditions will then be randomized to avoid potential biases linked to the sequence of conditions.

SUMMARY:
The purpose of this study is to investigate the cerebral activation during Classic Mirror Therapy (TMC) and especially during Virtual Mirror Therapy (TMV) in healthy subjects. It seems that the precuneus is involved in the effectiveness of mirror therapy. One goal of this study is to determine if there is a better activation of the precuneus during TMV than during TMC. Others goals are to compare cerebral activation during three different tasks (TMV, TMC and a simple motor task), to study the intra-subjects reproducibility of the measurement and the correlation between cerebral activation and feelings of the participants about the efficacity of the tasks.

DETAILED DESCRIPTION:
Mirror therapy is a rehabilitation technique that has been shown to be effective in restoring upper limb motor skills in patients with stroke. However, it comes up against certain constraints of clinical use such as installation difficulties or the obligation of symmetrical bilateral work. These constraints can be limited by the use of so-called 2nd generation virtual mirror therapy technologies. It is therefore likely that these new technologies will improve the feasibility and effectiveness of mirror therapy in rehabilitation. While the brain mechanisms involved in mirror therapy are not yet fully understood, the involvement of the precuneus has been demonstrated by a booming imaging method: fNIRS (functional Near Infra Red Spectroscopy). This method allows (like fMRI) to study cerebral neurovascular coupling. It is based on the fact that an activated region of the brain increases its local blood flow. Oxygenated hemoglobin (HbO) and deoxygenated (HbR) absorb infrared light and it is then possible to identify the cortical regions of the brain involved in a given task. This technique therefore makes it possible to study brain activation under more ecological conditions than fMRI and is therefore particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using a fNIRS apparatus, the brain regions involved in the performance of a classic mirror therapy task and a virtual mirror therapy task with the IVS3 (Intensive Visual Simulation) apparatus (Dessintey Technology).

The investigations will be carried out by the principal investigator or by specialized technicians from the neurology functional exploration department.

Each acquisition has a duration of 620 seconds, it begins with a rest period of 120 seconds, which corresponds to the baseline.

For each condition the movements are performed at a frequency of 0.5 Hz which seems to be the optimal frequency for observing cortical activation using a metronome. Each movement is therefore performed 10 times per block.

The order of placing the various conditions will be balanced. Between periods of movement, the subject is in a resting position for 30 seconds.

The "movement" and "rest" instructions are given at the start of each phase. The entire test will be repeated one week apart to assess the reproducibility of the measurements in healthy subjects.

The protocol has 3 conditions:

* A virtual TM task (TMV)
* A classic TM task (TMC)
* A control task (TC) Healthy subjects participating in the study will have two different acquisition times, each comprising 3 conditions.

After recruiting the subjects, the study investigator will check the inclusion and non-inclusion criteria.

If the subject can integrate the protocol, the two acquisition stages will then be scheduled one week apart.

On the day of the first acquisition, the subject will present to the neurology department at the time of his appointment.

The order of the 3 conditions will then be randomized to avoid potential biases linked to the sequence of conditions.

Then the fNIRS acquisition headset (Brite 24) will be installed by a specialized technician and the procurement instructions will be given.

The acquisition under the 3 conditions is then carried out: TC1, TMC1, TMV1 with a rest time of 10 minutes between each condition.

The subject's feelings after the TMC and TMV conditions will be evaluated using the visual analogue scale (VAS). 0 corresponding to a zero feeling and 10 to a very important feeling. The subject will be explained that the feeling could correspond to tingling sensations, a desire to mobilize the hand which is behind the mirror, a "disturbing", "bizarre" sensation.

The helmet is only removed at the end of the 3 spots The subject returns a week later for the 2nd acquisition phase during which the same acquisitions as during the 1st meeting are carried out and then participation in the study is terminated.

There will therefore be 6 tests for each healthy subject.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 40
* Right handed
* No neurological disease

Exclusion Criteria:

* Known allergy to components of the fNIRS device: neoprene

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Compare the level of precuneus activation during conventional mirror therapy (TMC) and virtual mirror therapy (TMV) | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs device

SECONDARY OUTCOMES:
Compare the level of activation of the precuneus during TMC and TC. | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs device
Compare the level of precuneus activation during TMV and TC. | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Compare the level of activation of contralateral motor regions to visual feedback during TMC and TMV. | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Compare the level of activation of the contralateral motor regions to visual feedback during TMV and TC. | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Compare the level of activation of the contralateral motor regions to visual feedback during TMC and TC. | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Evaluate the reproducibility of measurements | Day 0
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Evaluate the reproducibility of measurements | Day 7
  Changes in the concentration of oxyhemoglobin and deoxyhemoglobin measured with fnirs (functional Near Infra Red Spectroscopy) device
Compare the cortical regions involved during the different mirror therapy tasks and the feelings of the subjects. | Day 0
  Visual Analog Scale (VAS), minimal score is 0 (worst score) maximal score is 10 (better score)

CONTACTS AND LOCATIONS:
Overall Officials: Julien BONNAL, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Bae SJ, Jang SH, Seo JP, Chang PH. The Optimal Speed for Cortical Activation of Passive Wrist Movements Performed by a Rehabilitation Robot: A Functional NIRS Study. Front Hum Neurosci. 2017 Apr 20;11:194. doi: 10.3389/fnhum.2017.00194. eCollection 2017. PMID 28473763
- [Background] Bai Z, Fong KNK, Zhang J, Hu Z. Cortical mapping of mirror visual feedback training for unilateral upper extremity: A functional near-infrared spectroscopy study. Brain Behav. 2020 Jan;10(1):e01489. doi: 10.1002/brb3.1489. Epub 2019 Dec 5. PMID 31805613
- [Background] Brunetti M, Morkisch N, Fritzsch C, Mehnert J, Steinbrink J, Niedeggen M, Dohle C. Potential determinants of efficacy of mirror therapy in stroke patients--A pilot study. Restor Neurol Neurosci. 2015;33(4):421-34. doi: 10.3233/RNN-140421. PMID 26409402
- [Background] Calautti C, Jones PS, Naccarato M, Sharma N, Day DJ, Bullmore ET, Warburton EA, Baron JC. The relationship between motor deficit and primary motor cortex hemispheric activation balance after stroke: longitudinal fMRI study. J Neurol Neurosurg Psychiatry. 2010 Jul;81(7):788-92. doi: 10.1136/jnnp.2009.190512. Epub 2010 Apr 14. PMID 20392975
- [Background] Chang CS, Lo YY, Chen CL, Lee HM, Chiang WC, Li PC. Alternative Motor Task-Based Pattern Training With a Digital Mirror Therapy System Enhances Sensorimotor Signal Rhythms Post-stroke. Front Neurol. 2019 Nov 22;10:1227. doi: 10.3389/fneur.2019.01227. eCollection 2019. PMID 31824406
- [Background] Darbois N, Guillaud A, Pinsault N. Do Robotics and Virtual Reality Add Real Progress to Mirror Therapy Rehabilitation? A Scoping Review. Rehabil Res Pract. 2018 Aug 19;2018:6412318. doi: 10.1155/2018/6412318. eCollection 2018. PMID 30210873
- [Background] Ferrari M, Quaresima V. A brief review on the history of human functional near-infrared spectroscopy (fNIRS) development and fields of application. Neuroimage. 2012 Nov 1;63(2):921-35. doi: 10.1016/j.neuroimage.2012.03.049. Epub 2012 Mar 28. PMID 22510258
- [Background] Giraux P, Sirigu A. Illusory movements of the paralyzed limb restore motor cortex activity. Neuroimage. 2003 Nov;20 Suppl 1:S107-11. doi: 10.1016/j.neuroimage.2003.09.024. PMID 14597303
- [Background] Harmsen WJ, Bussmann JB, Selles RW, Hurkmans HL, Ribbers GM. A Mirror Therapy-Based Action Observation Protocol to Improve Motor Learning After Stroke. Neurorehabil Neural Repair. 2015 Jul;29(6):509-16. doi: 10.1177/1545968314558598. Epub 2014 Nov 21. PMID 25416737
- [Background] Inagaki Y, Seki K, Makino H, Matsuo Y, Miyamoto T, Ikoma K. Exploring Hemodynamic Responses Using Mirror Visual Feedback With Electromyogram-Triggered Stimulation and Functional Near-Infrared Spectroscopy. Front Hum Neurosci. 2019 Feb 26;13:60. doi: 10.3389/fnhum.2019.00060. eCollection 2019. PMID 30863295
- [Background] Jihun Kim, Jaehyo Kim. Robot-assisted mirroring exercise as a physical therapy for hemiparesis rehabilitation. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:4243-4246. doi: 10.1109/EMBC.2017.8037793. PMID 29060834
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Lee HM, Li PC, Fan SC. Delayed mirror visual feedback presented using a novel mirror therapy system enhances cortical activation in healthy adults. J Neuroeng Rehabil. 2015 Jul 11;12:56. doi: 10.1186/s12984-015-0053-1. PMID 26160599
- [Background] Li YC, Wu CY, Hsieh YW, Lin KC, Yao G, Chen CL, Lee YY. The Priming Effects of Mirror Visual Feedback on Bilateral Task Practice: A Randomized Controlled Study. Occup Ther Int. 2019 Nov 26;2019:3180306. doi: 10.1155/2019/3180306. eCollection 2019. PMID 31824233
- [Derived] Bonnal J, Ozsancak C, Prieur F, Auzou P. Video mirror feedback induces more extensive brain activation compared to the mirror box: an fNIRS study in healthy adults. J Neuroeng Rehabil. 2024 May 14;21(1):78. doi: 10.1186/s12984-024-01374-1. PMID 38745322